CLINICAL TRIAL: NCT03114423
Title: The Efficiency of Eye Movement Desensitization and Reprocessing (EMDR) for the Treatment of Substance Use Disorders: A Randomized Controlled Trial
Brief Title: Eye Movement Desensitization and Reprocessing (EMDR) as a Treatment of Substance Use Disorders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Center of Integrative Addiction Research, Austria (Other)
Collaborators: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMDR_1
Record Dates: First submitted 2017-04-11; First posted 2017-04-14 (Actual); Last update posted 2019-08-05 (Actual); Status verified 2019-08

CONDITIONS: Psychotherapy; Substance Use Disorders
Keywords: EMDR; Psychotherapy; Substance Use Disorders; Eye Movement Desensitization and Reprocessing
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment As Usual + Treatment with EMDR (Experimental)
  Interventions: Other: EMDR-Therapy
- Treatment As Usual + Cognitive Training (Sham Comparator)
  Interventions: Other: Sham Intervention

INTERVENTIONS:
Other: EMDR-Therapy — The EMDR-protocol from Hase (2008) was used
  Arms: Treatment As Usual + Treatment with EMDR
Other: Sham Intervention — For the training the COGPACK-program from Marker (2008) was used
  Arms: Treatment As Usual + Cognitive Training

SUMMARY:
The purpose of this clinical study is to examine the established, therapeutic EMDR intervention for patients with substance use disorders (SUD). The EMDR method is an integrative and structured therapeutic method which assumes that memories which have been dysfunctionally stored can lead to harmful behavior. The EMDR protocol used for this clinical trials has been specifically developed for patients with SUD - the results should be compared with traditional therapy. For the assessment of the EMDR treatment some questionnaires are given at several times.

DETAILED DESCRIPTION:
Substance use disorders (SUD) have been prominently described on a neuronal level as a chronic and relapsing brain disorder, which is associated with changes in emotion, motivation and cognition. Furthermore on a behavioral level, SUD have been found to be linked to an increased amount of attachment and personality pathology. More in general, SUD treatment has been demonstrated to be a complex phenomenon, with high relapse rates of 30-50% after (successful) treatment.

As emotion regulation is associated with a vast amount of parameters of mental health and psychological well-being such as more satisfied employment, healthier relationships, better academic performance, and physical health, the long-term abuse of drugs on the other hand plays a detrimental role in patients' emotions and mind-sets. Research suggests that individuals who cannot regulate their emotions in an adequate way in everyday life, experience more mental turbulences or confusions. In turn this deficit might lead to substance abuse as one kind of dysfunctional method to regulate inner tensions.

Specifically, an increased amount of impulsivity has been named as being predictive for addictive diseases. Accordingly, impulsivity was observed as being linked to a poorer SUD treatment outcome, especially by promoting relapse, as the emotion regulation is hindered and damaged in SUD patients. Thus the increase of capacities to moderate emotional strain becomes an important factor for the treatment of SUD. Accordingly, many SUD treatment approaches have developed specific techniques in order to address the deficient emotion regulation system. Furthermore a history of traumatic experiences may be essential for the therapeutic work, because individuals with SUD often present a history of trauma with comorbid rates of up to 75%. Consequentely, various findings suggest that traumatic experiences represent a high risk factor for the development of SUD.

The method of Eye Movement Desensitization and Reprocessing (EMDR) is an integrative and well structured psychotherapeutic treatment which has received approval as an efficacious evidence-based approach for posttraumatic stress disorder (PTSD). EMDR, as a psychotherapeutic technique, accelerates the accessing and reprocessing of traumatic materials and supports the brain to release the nervous system from these traumatic experiences by means of normal handling of emotional information. Due to the fact that up to 40% of individuals with PTSD turn to substance abuse in their lifetime, EMDR is effective in the treatment of SUD especially in case of unsolved traumata, which are keeping up the vicious circle of SUD. Furthermore several studies suggest that EMDR is effective in addiction treatment by significantly reducing substance craving and thus also the rate of relapse, extending consecutive sobriety, as well as more than twice as many graduates in EMDR integrated programs. However, the evidence of the efficacy and effectiveness of EMDR on addiction treatment is still limited, because many findings are preliminary as being narratively or just case-study based or paying less attention to the role of emotions. Therefore, the purpose of this study is to further explore and determine the effectiveness of EMDR for the regulation of emotional processes in long-term addiction treatment.

This study is conceptualized as a randomized controlled trial with two groups: EMDR + TAU vs. TAU + sham intervention (TAU: Treatment As Usual; the sham intervention is a cognitive training). The groups are compared pre-treatment, post-treatment, and there are two follow-up points of assessment: one month after post-treatment and three months after post-treatment. There will be a total sample of 60 clinical SUD male participants, which will be investigated during their in-patient stay at a therapeutic community center (after an initial phase of acclimatization of six weeks). One half of the sample: 30 participants will receive EMDR + TAU (experimental group; EG), the other half receives TAU + sham intervention (control group; CG).

ELIGIBILITY:
Inclusion Criteria:

* male
* SUD diagnosis
* age between 18 and 60 years
* patient must be stationary for at least six weeks
* patient must be full contractual capability

Exclusion Criteria:

* psychotic episode
* comorbid severe dissociative symptoms
* comorbid severe personality disorders
* organic conditional seizure disorders, and somatic disorders (e.g., severe cardiac arrhythmias).

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-04-07 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Emotion Regulation Questionnaire (ERQ) | Change of baseline values in ERQ after three treatments; follow-up_1 four weeks and follow-up_2 12 weeks after treatment.
  Emotion regulation is captured via 10 items on a 7-pint rating scale.

CONTACTS AND LOCATIONS:
Overall Officials: Human-Friedrich Unterrainer, PD DDr., Principal Investigator — Center of Integrative Addiction Research, Austria
Locations (1):
- Grüner Kreis, Verein zur Rehabilitation und Integration suchtkranker Menschen, Johnsdorf, Styria, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abel, N. J., & O'Brien, J. M. (2010). EMDR Treatment of Comorbid PTSD and Alcohol Dependence: A Case Example. Journal of EMDR Practice and Research, 4(2), 50-59. http://doi.org/10.1891/1933-3196.4.2.50.
- [Background] Abler, B., & Kessler, H. (2009). Emotion Regulation Questionnaire - Eine Deutschsprachige Fassung des ERQ von Gross und John. Diagnostica, 55(3), 144-152. http://doi.org/10.1026/0012-1924.55.3.144.
- [Background] Aldao A, Nolen-Hoeksema S, Schweizer S. Emotion-regulation strategies across psychopathology: A meta-analytic review. Clin Psychol Rev. 2010 Mar;30(2):217-37. doi: 10.1016/j.cpr.2009.11.004. Epub 2009 Nov 20. PMID 20015584
- [Background] Ursano RJ, Bell C, Eth S, Friedman M, Norwood A, Pfefferbaum B, Pynoos JD, Zatzick DF, Benedek DM, McIntyre JS, Charles SC, Altshuler K, Cook I, Cross CD, Mellman L, Moench LA, Norquist G, Twemlow SW, Woods S, Yager J; Work Group on ASD and PTSD; Steering Committee on Practice Guidelines. Practice guideline for the treatment of patients with acute stress disorder and posttraumatic stress disorder. Am J Psychiatry. 2004 Nov;161(11 Suppl):3-31. No abstract available. PMID 15617511
- [Background] Brown, S. H., Gilman, S. G., Goodman, E. G., Adler-Tapia, R., & Freng, S. (2015). Integrated Trauma Treatment in Drug Court: Combining EMDR Therapy and Seeking Safety. Journal of EMDR Practice and Research, 9(3), 123-136. http://dx.doi.org/10.1891/1933-3196.9.3.123
- [Background] Ersche KD, Sahakian BJ. The neuropsychology of amphetamine and opiate dependence: implications for treatment. Neuropsychol Rev. 2007 Sep;17(3):317-36. doi: 10.1007/s11065-007-9033-y. Epub 2007 Aug 10. PMID 17690986
- [Background] Flores, J. P., 2004. Addiction as an Attachment Disorder. Maryland: Jason Aronson Inc. Publishers. Franke, G. H. (2000). Brief Symptom Inventory (BSI). Göttingen: Beltz.
- [Background] Hase, M., Schallmayer, S., & Sack, M. (2008). EMDR Reprocessing of the Addiction Memory: Pretreatment, Posttreatment, and 1-Month Follow-Up. Journal of EMDR Practice and Research, 2(3), 170-179. http://doi.org/10.1891/1933-3196.2.3.170.
- [Background] Homer BD, Solomon TM, Moeller RW, Mascia A, DeRaleau L, Halkitis PN. Methamphetamine abuse and impairment of social functioning: a review of the underlying neurophysiological causes and behavioral implications. Psychol Bull. 2008 Mar;134(2):301-10. doi: 10.1037/0033-2909.134.2.301. PMID 18298273
- [Background] Jacobsen LK, Southwick SM, Kosten TR. Substance use disorders in patients with posttraumatic stress disorder: a review of the literature. Am J Psychiatry. 2001 Aug;158(8):1184-90. doi: 10.1176/appi.ajp.158.8.1184. PMID 11481147
- [Background] Klinitzke G, Romppel M, Hauser W, Brahler E, Glaesmer H. [The German Version of the Childhood Trauma Questionnaire (CTQ): psychometric characteristics in a representative sample of the general population]. Psychother Psychosom Med Psychol. 2012 Feb;62(2):47-51. doi: 10.1055/s-0031-1295495. Epub 2011 Dec 27. German. PMID 22203470
- [Background] Lee, C. W., Taylor, G., & Drummond, P. D. (2006). The active ingredient in EMDR: Is it traditional exposure or dual focus of attention? Clinical Psychology and Psychotherapy, 13(2), 97-107. http://doi.org/10.1002/cpp.479.
- [Background] Loree AM, Lundahl LH, Ledgerwood DM. Impulsivity as a predictor of treatment outcome in substance use disorders: review and synthesis. Drug Alcohol Rev. 2015 Mar;34(2):119-34. doi: 10.1111/dar.12132. Epub 2014 Mar 31. PMID 24684591
- [Background] Marich J. Eye movement desensitization and reprocessing in addiction continuing care: a phenomenological study of women in recovery. Psychol Addict Behav. 2010 Sep;24(3):498-507. doi: 10.1037/a0018574. PMID 20853935
- [Background] Marissen MA, Franken IH, Blanken P, van den Brink W, Hendriks VM. Cue exposure therapy for the treatment of opiate addiction: results of a randomized controlled clinical trial. Psychother Psychosom. 2007;76(2):97-105. doi: 10.1159/000097968. PMID 17230050
- [Background] Meysami-Bonab, S., Abolghasemi, A., Sheikhian, M., Barahmand, U., & Rasooliazad, M. (2012). The Effectiveness of Eye Movement Desensitization and Reprocessing Therapy on the Emotion Regulation and Emotion Recognition of Addicted Individuals. Zahedan Journal of Research in Medical Sciences, 14(10), 33-37.
- [Background] Moos RH, Moos BS. Rates and predictors of relapse after natural and treated remission from alcohol use disorders. Addiction. 2006 Feb;101(2):212-22. doi: 10.1111/j.1360-0443.2006.01310.x. PMID 16445550
- [Background] Ouimette P, Coolhart D, Funderburk JS, Wade M, Brown PJ. Precipitants of first substance use in recently abstinent substance use disorder patients with PTSD. Addict Behav. 2007 Aug;32(8):1719-27. doi: 10.1016/j.addbeh.2006.11.020. Epub 2006 Dec 22. PMID 17188816
- [Background] Parker, J. D. A., Taylor, R. N., Eastabrook, J. M., Schell, S. L., & Wood, L. M. (2008). Problem gambling in adolescence: Relationships with internet misuse, gaming abuse and emotional intelligence. Personality and Individual Differences, 45(2), 174-180. http://doi.org/10.1016/j.paid.2008.03.018
- [Background] Schmidt S, Strauss B, Hoger D, Brahler E. [The Adult Attachment Scale (AAS) - psychometric evaluation and normation of the German version]. Psychother Psychosom Med Psychol. 2004 Sep-Oct;54(9-10):375-82. doi: 10.1055/s-2003-815000. German. PMID 15343479
- [Background] Schulz, H., Lang, K., Nübling, R., & Koch, U. (2003). Psychometrische Überprüfung einer Kurzform des Fragebogens zur Psychotherapiemotivation - FPTM-23. Diagnostica, 49(2), 83-93. http://doi.org/10.1026//0012-1924.49.2.83
- [Background] Solomon, R., & Shapiro, F. (2008). EMDR and the adaptive information processing model: Potential mechanisms of change. Journal of EMDR Practice and Research, 2(4), 315-325. http://doi.org/10.1891/1933-3196.2.4.315
- [Background] Swendsen J, Conway KP, Degenhardt L, Glantz M, Jin R, Merikangas KR, Sampson N, Kessler RC. Mental disorders as risk factors for substance use, abuse and dependence: results from the 10-year follow-up of the National Comorbidity Survey. Addiction. 2010 Jun;105(6):1117-28. doi: 10.1111/j.1360-0443.2010.02902.x. Epub 2010 Mar 10. PMID 20331554
- [Background] Torchalla I, Nosen L, Rostam H, Allen P. Integrated treatment programs for individuals with concurrent substance use disorders and trauma experiences: a systematic review and meta-analysis. J Subst Abuse Treat. 2012 Jan;42(1):65-77. doi: 10.1016/j.jsat.2011.09.001. Epub 2011 Oct 27. PMID 22035700
- [Background] Trinidad, D. R., Unger, J. B., Chou, C. P., & Anderson Johnson, C. (2004). The protective association of emotional intelligence with psychosocial smoking risk factors for adolescents. Personality and Individual Differences, 36(4), 945-954. http://doi.org/10.1016/S0191-8869(03)00163-6
- [Background] Verdejo-Garcia A, Lawrence AJ, Clark L. Impulsivity as a vulnerability marker for substance-use disorders: review of findings from high-risk research, problem gamblers and genetic association studies. Neurosci Biobehav Rev. 2008;32(4):777-810. doi: 10.1016/j.neubiorev.2007.11.003. Epub 2008 Jan 17. PMID 18295884
- [Background] Verdejo-Garcia A, Lopez-Torrecillas F, Gimenez CO, Perez-Garcia M. Clinical implications and methodological challenges in the study of the neuropsychological correlates of cannabis, stimulant, and opioid abuse. Neuropsychol Rev. 2004 Mar;14(1):1-41. doi: 10.1023/b:nerv.0000026647.71528.83. PMID 15260137
- [Background] Xie H, McHugo GJ, Fox MB, Drake RE. Substance abuse relapse in a ten-year prospective follow-up of clients with mental and substance use disorders. Psychiatr Serv. 2005 Oct;56(10):1282-7. doi: 10.1176/appi.ps.56.10.1282. PMID 16215196